CLINICAL TRIAL: NCT01280617
Title: Low Dose Thymoglobulin As Induction Agent on Prednisone-Free Regimens of Renal Transplant Recipients
Brief Title: Low Dose Thymoglobin in Renal Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahey Clinic (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-065
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Acute Renal Failure
Keywords: Renal Transplant; Thymoglubulin
MeSH Terms: conditions — Acute Kidney Injury | interventions — thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thymoglobulin 1.25mg/kg dose (Experimental): The safety and efficacy of low dose Thymoglobulin (1.25mg/kg) as an induction agent in renal transplant subjects.
  Interventions: Drug: Thymoglobulin
- Thymoglobulin 0.75mg/kg dose (Experimental): The safety and efficacy of low dose Thymoglobulin (0.75mg/kg) as an induction agent in renal transplant subjects.
  Interventions: Drug: Thymoglobulin 0.75mg/kg dose

INTERVENTIONS:
Drug: Thymoglobulin — Thymoglobulin 1.25mg/kg dose
  Arms: Thymoglobulin 1.25mg/kg dose
Drug: Thymoglobulin 0.75mg/kg dose — Thymoglobulin
  Other Names: Thymoglobulin
  Arms: Thymoglobulin 0.75mg/kg dose

SUMMARY:
This is a planned single center prospective randomized study evaluating the safety and efficacy of low dose thymoglobulin as induction agent in renal transplant recipients. Inclusion criteria will be adult renal transplant recipients who are not sensitized against their potential donors. The patients who agree to participate in the study will be randomly assigned to either thymoglobulin at 1.25mg/kg x 3 doses or 0.75mg/kg x 3 doses. There will be 86 sealed envelopes to perform the randomization process. 43 envelopes with 1.25mg/kg dosing and the other 43 envelopes with 0.75mg/kg dosing. The investigators will sequentially choose the sealed envelopes at the time of the patient randomization process. All patients will be started on our standard immunosupression regimen of prograf/cellcept and a fast steroid taper. Data will be obtained from every patient for up to one year post-transplant.

DETAILED DESCRIPTION:
Detailed Study Design:

This is a planned single center prospective randomized study evaluating the safety and efficacy of low dose thymoglobulin as induction agent in renal transplant recipients. Inclusion criteria will be adult renal transplant recipients who are not sensitized against their potential donors. The patients who agree to participate in the study will be randomly assigned to either thymoglobulin at 1.25mg/kg x 3 doses or 0.75mg/kg x 3 doses. There will be 86 sealed envelopes to perform the randomization process. 43 envelopes with 1.25mg/kg dosing and the other 43 envelopes with 0.75mg/kg dosing. The investigators will sequentially choose the sealed envelopes at the time of the patient randomization process. All patients will be started on our standard immunosupression regimen of prograf/cellcept and a fast steroid taper. Data will be obtained from every patient for up to one year post-transplant.

The investigators will obtain the following information at the time of consent:

1. Type of renal transplant (living vs cadaveric)
2. HLA matching
3. CMV status of donor and recipient
4. EBV status of donor and recipient
5. Creatinine prior to transplantation
6. Urinalysis at the time of transplantation
7. Primary renal disease
8. Weight of the renal transplant
9. BMI of the recipient and donor
10. Age of the donor and recipient
11. Sex of the donor and recipient
12. White blood cell count
13. Hemoglobin
14. Platelets
15. History of infections
16. History of malignancies

During each of the clinic visits the investigators will obtain the following information:

1. Creatinine
2. Urinalysis
3. White blood cell count
4. Hemoglobin
5. Platelets
6. Weight of the recipient
7. Infections
8. Malignancies
9. Renal biopsy report if a biopsy was performed

In addition to the standard of care laboratories, the investigators will ask patients to give us 7 additional green tubes, one purple tube and two red tubes which will be drawn at the time of standard of care laboratories pre-transplantation, 3 months post-transplant, 6 months post-transplant and 12 months post-transplant. This tubes will be used to measure CD4, CD8, CD19, CD20, CD68 cells as these are cells that are believed to be affected by the use of thymoglobulin.

If the patient is to have a renal transplant biopsy at any time during the 12 months of the study, any excess tissue may be utilized for staining of special cell markers including CD4, CD8, CD19, CD20 and CD68.

Subject inclusion criteria: Potential adult renal transplant recipients

Subject exclusion criteria: Sensitized renal transplant recipients

Methods of statistical analysis to be employed in preparation of reports:

The investigators are planning a study with 1 control per experimental subject, an accrual interval of 24 time units, and additional follow-up after the accrual interval of 12 time units. In a previous study the median survival time on the control treatment was 36 time units. If the true hazard ratio (relative risk) of control subjects relative to experimental subjects is 5, the investigators will need to study 43 experimental subjects and 43 control subjects to be able to reject the null hypothesis that the experimental and control survival curves are equal with probability (power) .800. The Type I error probability associated with this test of this null hypothesis is 0.05. T-tests will be used to compare both groups.

Thymoglobulin (rabbit antithymocyte globulin) is FDA approved for the treatment of acute cellular rejection. Nevertheless, for at least the past 10 years this medication has been utilized as induction agent in renal transplant recipients. This is because an induction agent allows prednisone withdrawal in renal transplant recipients.

Prednisone withdrawal is extremely important in renal transplant recipients as old protocols that allowed long term prednisone use compromised the long term health of renal transplant recipients. Not only does prednisone increase markedly the risk of development of diabetes and osteoporosis, but is also increases drastically the risk of fractures, which is a very common cause of mortality in long term prednisone renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

Potential Adult Renal Transplant Patients -

Exclusion Criteria:

Sensitized Renal Transplant Patients

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-10; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simpson, Principal Investigator — Lahey Hospital & Medical Ctr
Locations (1):
- Lahey Clinic, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grafals M, Smith B, Murakami N, Trabucco A, Hamill K, Marangos E, Gilligan H, Pomfret EA, Pomposelli JJ, Simpson MA, Azzi J, Najafian N, Riella LV. Immunophenotyping and efficacy of low dose ATG in non-sensitized kidney recipients undergoing early steroid withdrawal: a randomized pilot study. PLoS One. 2014 Aug 11;9(8):e104408. doi: 10.1371/journal.pone.0104408. eCollection 2014. PMID 25111080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All unsensitized renal transplant recipients were considered eligible and were approached for consent. Inclusion dates were October 2010 until April 2013. A total of 58 patients were approached; 44 consented and were enrolled in the protocol
Period: Overall Study
Arm/Group | Thymoglobulin 1.25mg/kg Dose | Thymoglobulin 0.75mg/kg Dose
Started | 23 | 21
Completed | 23 | 20
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thymoglobulin 1.25mg/kg Dose | Thymoglobulin 0.75mg/kg Dose | Total
Number analyzed (Participants) | 23 | 20 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 17 | 40
  >=65 years | 0 | 3 | 3
Sex/Gender, Customized [Count of Participants; unit: Participants]
  males | 16 | 16 | 32
  females | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Rates of Acute Cellular Rejection Between Study Group
Description: Incidence of Biopsy Proven Acute Rejection at 1 year post transplant:
Time Frame: 1 year from date of transplant
Measure: Number; unit: Number of rejection
Groups:
- Thymoglobulin 1.25mg/kg Dose: Thymoglobulin 1.25mg/kg dose All Cause mortality 0/23
- Thymoglobulin 0.75mg/kg Dose: Thymoglobulin 0.75mg/kg dose All Cause Mortality 3/20 - 2 with pre-existing cardiac disease, diabetes, and history of smoking
Arm/Group | Thymoglobulin 1.25mg/kg Dose | Thymoglobulin 0.75mg/kg Dose
Number analyzed (Participants) | 23 | 20
Number of rejection | 4 | 2
Statistical Analysis 1: Comparison: Thymoglobulin 1.25mg/kg Dose vs Thymoglobulin 0.75mg/kg Dose; Test type: Superiority; p < 0.05, t-test, 2 sided; Continuous variables analyzed using 2-tailed t test or Mann Whitney tes.. Categorical variables analyzed using Chi-Square or Fisher's Exact test
Statistical Analysis 2: Comparison: Thymoglobulin 1.25mg/kg Dose vs Thymoglobulin 0.75mg/kg Dose; Test type: Superiority; p < 0.05, t-test, 2 sided

2. Secondary Outcome: , "Total Number of Adverse Events, Including Any Infections, Leucopenia, and Malignancy"
Description: Number of individual adverse events in high versus low dose Thymoglobulin groups will be tabulated and statistical analyses performed
Time Frame: 1 year from date of transplant
Measure: Number; unit: Adverse Events
Arm/Group | Thymoglobulin 1.25mg/kg Dose | Thymoglobulin 0.75mg/kg Dose
Number analyzed (Participants) | 23 | 20
Adverse Events | 3 | 8

ADVERSE EVENTS:
Time Frame: Day of kidney transplant until end of first post transplant year
Arm/Group | Thymoglobulin 1.25mg/kg Dose | Thymoglobulin 0.75mg/kg Dose
All-Cause Mortality (participants affected / at risk) | 0/23 | 3/20
Serious Adverse Events (participants affected / at risk) | 3/23 | 2/20
Other Adverse Events (participants affected / at risk) | 3/23 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thymoglobulin 1.25mg/kg Dose (N=23) | Thymoglobulin 0.75mg/kg Dose (N=20)
Serious Infections (Infections and infestations) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thymoglobulin 1.25mg/kg Dose (N=23) | Thymoglobulin 0.75mg/kg Dose (N=20)
Delayed Graft Function (Renal and urinary disorders) | 3 (3) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No